CLINICAL TRIAL: NCT05250024
Title: Cranioplasty Using Patient Specific Implants Polyether Ether Ketone Versus Ultra-High Molecular Weight Polyethylene: A Randomized Controlled Trial
Brief Title: Synthetic Cranioplasty PEEK Versus UHMWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam SK Abdelwahed, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRANIOPEEK/UHMWP
Record Dates: First submitted 2022-01-31; First posted 2022-02-22 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Cranium; Deformity
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- UHMWP Cranioplasty (Experimental): synthetic reconstruction of cranial defects using computer guided milled UHMWP implants
  Interventions: Device: UHMWP Cranioplasty
- PEEK Cranioplasty (Active Comparator): synthetic reconstruction of cranial defects using computer guided milled PEEK
  Interventions: Device: PEEK Cranioplasty

INTERVENTIONS:
Device: UHMWP Cranioplasty — patient specific cranial implant
  Arms: UHMWP Cranioplasty
Device: PEEK Cranioplasty — patient specific cranial implant
  Arms: PEEK Cranioplasty

SUMMARY:
The purpose of this study is to report the investigators experience with synthetic reconstruction of cranial defects using computer guided milled UHMWP, in terms of benefits and limitations both clinically and radiographically in comparison to PEEK implants.

DETAILED DESCRIPTION:
Statement of the problem:

To this date, there is still no consensus on the ideal material for cranial reconstruction. Research journey involved the use of autologous grafts, allografts, xenografts, and a wide array of synthetic materials for cranioplasty. The autologous bone flap, although associated with less infection than allo or xenografts, is not always a possibility after comminution or osteomyelitis and still has the common drawbacks of storage, aseptic bone flap necrosis (ABFR) and the need for a second surgery. Titanium offers lower cost but is quite difficult to shape, radiopaque and exhibits high dehiscence with thin skin biotypes. Polyetheretherketone (PEEK) has been gaining popularity during the recent years for lower rates of graft failure, however, it still holds a risk of postoperative inflammatory complications, is of exceedingly high cost most studies utilizing it are retrospective and observational.

Rationale for conducting the research:

Cranioplasty procedures carry functional and esthetic challenges and the most suitable graft to be used remains controversial. UHMWP use in biomedical applications is greatly due to its outstanding mechanical properties and biocompatibility which, when coupled with three D computer guided milling technology to reconstruct complex and large cranial defects, can provide durable patient specific implants (PSI). However, no interventional studies exist in the literature on its application in cranioplasty.

Explanation for choice of comparators:

PEEK as a semicrystalline thermoplastic polymer has a thickness and elasticity comparable to cortical bone making it one of the most commonly used bone substitute materials and is currently recommended as a standard viable option for cranial defects.

ELIGIBILITY:
Inclusion Criteria:

* Cranial defect patients
* Patients eligible for simultaneous craniectomy and cranioplasty.
* ASA I & II

Exclusion Criteria:

* Active infection.
* Medically compromised patients (ASA ≥3).
* Hydrocephalus/Brain Swelling

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Cosmetic patient satisfaction | 6 months
  Method: Questionnaire, Satisfaction Scale [ 1 Dissatisfied - 5 Highly satisfied ]

SECONDARY OUTCOMES:
Overall complications | 6 months
  Method: Clinical exam, Unit: Binary Y/N
implant failure | 6 months
  Method: Clinical exam, Unit: Binary Y/N

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh A Sayed, Professor, Study Director — Cairo University
Locations (1):
- Nasser Institute Hospital, Cairo, Shubra, Egypt